CLINICAL TRIAL: NCT04234750
Title: The Evaluation of the Safety and Effectiveness of Mesenchymal Stem Cell-derived Pleiotropic Factor in the Treatment of Donor Sites
Brief Title: Mesenchymal Stem Cell-derived Pleiotropic Factor in the Treatment of Donor Sites
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xiaobing Fu, Proffessor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-02
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Evaluate the Safety and Effectiveness of Mesenchymal Stem Cell Conditioned Medium-derived Pleiotropic Factor in Treating Donor Sites

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no intervention
- experimental group (Experimental): mesenchymal stem cell conditioned medium-derived pleiotropic factor
  Interventions: Biological: mesenchymal stem cell conditioned medium-derived pleiotropic factor

INTERVENTIONS:
Biological: mesenchymal stem cell conditioned medium-derived pleiotropic factor — After the patient is enrolled, when the patient's condition is stable, he is ready to undergo skin transplantation. For the donor site, an electric dermatome was used to remove the skin. The two donor areas of the same patient were divided into a pleiotropic factor group and a blank group randomly. After placing a coarse mesh vaseline oil gauze, then cover a certain thickness of sterile gauze and pressure bandage.
  Arms: experimental group

SUMMARY:
Skin grafting is a standard treatment for deep wounds, but care of the donor site after transplantation is very important. The means of accelerating wound healing can increase overall patient satisfaction. In recent years, cytokine therapy has been an important strategy to promote tissue repair.Mesenchymal stem cells (MSC) have been considered the star cells that promote tissue repair. It works mainly through paracrine. Many biological effectors, including IGF-1, vascular endothelial growth factor (VEGF), TGF-β1, and hepatocyte growth factor (HGF), have been found and reported in various MSC conditioned media (MSC-CM), And play a role in promoting tissue repair and regeneration. In here, we aim to explore the MSC-CM-derived pleiotropic factor in treating donor sites and further evaluate its safety and effectiveness

ELIGIBILITY:
Inclusion Criteria:

Mainly mild to moderate burns, III ° burn area is less than 20% (trauma factor is thermal burn); Thick-thickness skin (thickness 0.2-0.3mm), donor area and medium-thickness skin (thick 0.3-0.5mm) for the skin area study separately; Psychologically stable and able to complete the test process-

Exclusion Criteria:

History of clotting disorders, uncontrolled diabetes; Drug abuse, excessive drinking, malignant or autoimmune diseases, chemotherapy and immunosuppressive therapy; Significant local infection or combined systemic infection; Patients with severe heart, lung, liver, kidney, blood system and mental and nervous system diseases; Women during pregnancy and lactation-

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
wound healing rate | 1 month
  Original wound area minus unhealed wound area divided by original wound area

SECONDARY OUTCOMES:
Vancouver score | 6 months
  Score according to scale

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobing Fu, doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- People's Liberation Army Central Air Force Hospital, Datong, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Need to contact the researcher and open sharing after the researcher's consent
Supporting Information: Study Protocol
Time Frame: One year after clinical trial
Access Criteria: The way of sharing IPD has not yet been determined